CLINICAL TRIAL: NCT00260117
Title: Long-Term Exercise Maintenance Via Internet Support
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Paul T. Williams, Lawrence Berkeley Laboratory
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DK66738 (completed)
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2010-02

CONDITIONS: Obesity; Inactivity
Keywords: Exercise; Physical activity; walking; running
MeSH Terms: conditions — Obesity; Sedentary Behavior; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Exercise — Referal to a website

SUMMARY:
Each year, a significant portion of men and women who engage in physical activities such as walking or running reduce their activity and by doing so place themselves at greater risk of obesity, heart disease, and diabetes. Our own prospective epidemiological studies of runners and walkers suggest that during 7.6 years of follow-up over 40% have reduced their mileage by half or more. Research suggests that social support, perceived health benefits, resiliency to interruptions in training, and exercise self-efficacy predict successful maintenance. We have found that runners who successfully maintained or increased their running mileage during this follow-up were more likely to have participated in social events such as marathon, half-marathon, or 10km races.

The purpose of this study is to build upon our current Internet-based survey tools (www.healthsurvey.org) for tracking physical activity and nutrition on full-function activity and diet logs. The existing software allows participants to visualize their accumulated running and walking mileage on a virtual transcontinental route starting in Yorktown, Virginia and ending in Florence, Oregon. To the existing software, we will add the ability to: 1) choose named or anonymous running and walking partners with similar goals and abilities to travel with (or race against) along the transcontinental trail, 2) communicate with partners to provide mutual support, 3) compete as part of virtual running and walking teams created by the user, and 4) be recognized for completing each state on an awards page (optional). Interest in the site will be maintained by providing regular updates on scientific research on running and walking through our proprietary software. The updates will be created from PubMed abstracts that are made more reader friendly by defining all scientific terms in pop-up balloons.

DETAILED DESCRIPTION:
Participants are refered to a specially designed website to encourage participation

ELIGIBILITY:
Inclusion Criteria:

* Currently walking or running for exercise Prior participation in the National Runners' or Walkers' Health Studies

Exclusion Criteria:

* Under 18 years old No internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16000 (Estimated)
Dates: Start 2005-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Self-reported body weight | through2007

SECONDARY OUTCOMES:
Morbidity | Through 2007

CONTACTS AND LOCATIONS:
Overall Officials: Paul T Williams, PhD, Principal Investigator — Lawrence Berkeley National Laboratory
Locations (1):
- Lawrence Berkeley National Laboratory, Berkeley, California, United States